CLINICAL TRIAL: NCT04498273
Title: COVID-19 Outpatient Thrombosis Prevention Trial A Multi-center Adaptive Randomized Placebo-controlled Platform Trial Evaluating the Efficacy and Safety of Anti-thrombotic Strategies in COVID Adults Not Requiring Hospitalization at Time of Diagnosis
Brief Title: COVID-19 Positive Outpatient Thrombosis Prevention in Adults Aged 40-80
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: an event rate lower than anticipated
Sponsor: Frank C Sciurba (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Frank C Sciurba, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTIV4-Outpatient
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — apixaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Apixaban 2.5mg (Active Comparator): Anticoagulation: prophylactic dose Apixaban 2.5mg po bid
  Interventions: Drug: Apixaban 2.5 MG
- Apixaban 5mg (Active Comparator): Anticoagulation: therapeutic dose Apixaban 5.0mg po bid
  Interventions: Drug: Apixaban 5MG
- Aspirin (Active Comparator): Antiplatelet agent: low dose aspirin 81mg po qd
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban 2.5 MG — Subjects will be contacted either electronically or by telephone within 24 hours of randomization to confirm receipt of the study treatment. Study drug will be shipped to subjects home. Subjects will take Apixaban 2.5 MG twice a day; once in the morning and once in the evening for 45 days. Subjects will be contacted (electronic or telephone) minimally weekly after initial start of study medication and contact will continue up to day 75 after starting study treatment. Follow up electronic contact will be dependent on initial patient response, compliance with response, and medication adherence, for the trial duration using electronic contacts and through telephone contacts. Participants will be queried for any clinically relevant endpoints, especially major bleeding, or need to seek healthcare attention for any reason. Follow-up will occur from the time of study drug receipt and through the 30 day safety period.
  Arms: Apixaban 2.5mg
Drug: Apixaban 5MG — Subjects will be contacted either electronically or by telephone within 24 hours of randomization to confirm receipt of the study treatment. Study drug will be shipped to subjects home. Subjects will take Apixaban 5 MG twice a day; once in the morning and once in the evening for 45 days. Subjects will be contacted (electronic or telephone) minimally weekly after initial start of study medication and contact will continue up to day 75 after starting study treatment. Follow up electronic contact will be dependent on initial patient response, compliance with response, and medication adherence, for the trial duration using electronic contacts and through telephone contacts. Participants will be queried for any clinically relevant endpoints, especially major bleeding, or need to seek healthcare attention for any reason. Follow-up will occur from the time of study drug receipt and through the 30 day safety period.
  Arms: Apixaban 5mg
Drug: Aspirin — Subjects will be contacted either electronically or by telephone within 24 hours of randomization to confirm receipt of the study treatment. Study drug will be shipped to subjects home. Subjects will take Aspirin twice a day; once in the morning and once in the evening for 45 days. Subjects will be contacted (electronic or telephone) minimally weekly after initial start of study medication and contact will continue up to day 75 after starting study treatment. Follow up electronic contact will be dependent on initial patient response, compliance with response, and medication adherence, for the trial duration using electronic contacts and through telephone contacts. Participants will be queried for any clinically relevant endpoints, especially major bleeding, or need to seek healthcare attention for any reason. Follow-up will occur from the time of study drug receipt and through the 30 day safety period.
  Arms: Aspirin
Drug: Placebo — Subjects will be contacted either electronically or by telephone within 24 hours of randomization to confirm receipt of the study treatment. Study placebo will be shipped to subjects home. Subjects will take placebo twice a day; once in the morning and once in the evening for 45 days. Subjects will be contacted (electronic or telephone) minimally weekly after initial start of study medication and contact will continue up to day 75 after starting study treatment. Follow up electronic contact will be dependent on initial patient response, compliance with response, and medication adherence, for the trial duration using electronic contacts and through telephone contacts. Participants will be queried for any clinically relevant endpoints, especially major bleeding, or need to seek healthcare attention for any reason. Follow-up will occur from the time of study drug receipt and through the 30 day safety period.
  Arms: Placebo

SUMMARY:
A multi-center adaptive randomized placebo-controlled platform trial evaluating the efficacy and safety of anti-thrombotic strategies in COVID-19 adults not requiring hospitalization at time of diagnosis

DETAILED DESCRIPTION:
The COVID-19 Outpatient Thrombosis Prevention Trial is a multi-center adaptive randomized double-blind placebo-controlled platform trial to compare the effectiveness of anti-coagulation with anti-platelet agents and with placebo to prevent thrombotic events in patients diagnosed with COVID-19 who have evidence of increased inflammation based on elevated D-dimer and hsCRP levels, yet are not admitted to hospital as COVID-19 related symptoms are currently stable. Participants will all be adults between 40 and 79 years who will be enrolled from approximately 100 facilities, such as emergency rooms and other settings where a physician is present to evaluate the patient for inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion:

* COVID-19+ in past 14 days
* Platelets > 100,000
* eGFR > 30ml/min

Exclusion:

* Hospitalized
* Contradiction/ other indication for anti-coagulation
* Pregnancy
* Active cancer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sciurba, Principal Investigator — University of Pittsburgh
Locations (70):
- United States (70):
  - University of Southern California, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Zuckerberg San Francisco General, San Francisco, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Pine Ridge Family Medicine, Colorado Springs, Colorado
  - Life Tree Health, Inc., Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - University of Florida at Gainesville, Gainesville, Florida
  - Vital Pharma Research, Hialeah, Florida
  - Advanced Research for Health Improvement, LLC, Immokalee, Florida
  - University of Floridia at Jacksonville, Jacksonville, Florida
  - Lakeland Regional, Lakeland, Florida
  - Total Research Group LLC, Miami, Florida
  - Jackson Memorial, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Innovation Clinical Trials, Palmetto Bay, Florida
  - Bond Community Health Center, Tallahassee, Florida
  - Tallahassee Memorial, Tallahassee, Florida
  - USF Tampa General Hospital, Tampa, Florida
  - Alliance Clinical Research, Tampa, Florida
  - Hawaii Pacific Health, Honolulu, Hawaii
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - UIC - Mile Square, Chicago, Illinois
  - Jesse Brown VA, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Olivo Wellness Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Ascension Via Christi, Wichita, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Jadestone Clinical Research, LLC, Gaithersburg, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - GFC of Southeastern Michigan, Detroit, Michigan
  - SRI International, Plymouth, Michigan
  - Metro Health-University of Michigan Health, Wyoming, Michigan
  - Raritan Bay Primary Care and Cardiology Associates, Matawan, New Jersey
  - G&S Medical Associates, LLC, Paterson, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Strong Memorial, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Spinal Pain and Rehab Medicine, Yonkers, New York
  - Duke, Durham, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - The Heart and Medical Center, Durant, Oklahoma
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - UPMC Passavant Cranberry, Cranberry, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC East, Monroeville, Pennsylvania
  - UPMC Magee, Pittsburgh, Pennsylvania
  - UPMC Presby, Pittsburgh, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant McCandless, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Pharma Tex Research, Amarillo, Texas
  - Ascension Seton Medical Center, Austin, Texas
  - Baptist Beaumont, Beaumont, Texas
  - McGoven Medical School - UT- Houston, Houston, Texas
  - Diversifield Medical Practices, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Mesquite Regional Internal Medicine, Mesquite, Texas
  - University of Texas at Tyler, Tyler, Texas
  - University of Texas at Rio Grande Valley, Weslaco, Texas
  - Intermountain Healthcare, Murray, Utah
  - Community Care of Clay, Clay, West Virginia
  - University Healthcare Physicians, Harpers Ferry, West Virginia
  - Community Care of Weston, Weston, West Virginia
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Bledsoe J, Woller SC, Brooks M, Sciurba FC, Krishnan JA, Martin D, Hou P, Lin JY, Kindzelski A, Handberg E, Kirwan BA, Zaharris E, Castro L, Shapiro NL, Pepine CJ, Majercik S, Fu Z, Zhong Y, Venugopal V, Lai YH, Ridker PM, Connors JM. Clinically stable covid-19 patients presenting to acute unscheduled episodic care venues have increased risk of hospitalization: secondary analysis of a randomized control trial. BMC Infect Dis. 2023 May 15;23(1):325. doi: 10.1186/s12879-023-08295-9. PMID 37189091
- [Derived] Connors JM, Brooks MM, Sciurba FC, Krishnan JA, Bledsoe JR, Kindzelski A, Baucom AL, Kirwan BA, Eng H, Martin D, Zaharris E, Everett B, Castro L, Shapiro NL, Lin JY, Hou PC, Pepine CJ, Handberg E, Haight DO, Wilson JW, Majercik S, Fu Z, Zhong Y, Venugopal V, Beach S, Wisniewski S, Ridker PM; ACTIV-4B Investigators. Effect of Antithrombotic Therapy on Clinical Outcomes in Outpatients With Clinically Stable Symptomatic COVID-19: The ACTIV-4B Randomized Clinical Trial. JAMA. 2021 Nov 2;326(17):1703-1712. doi: 10.1001/jama.2021.17272. PMID 34633405
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from a variety of different facilities where (a) a clinician can evaluate the patient for inclusion and exclusion criteria, and (b) where blood samples can be arranged to be sent for D-dimer, hsCRP, calculated creatinine clearance, and platelet count. COVID-19 testing needs to be confirmed positive within the past 14 days. Serum or urine pregnancy test results will be required for women of childbearing potential before starting study treatment.
Groups:
- Asprin: Antiplatelet agent: low dose aspirin 81mg po qd
- Placebo: Only Placebo
Period: Overall Study
Arm/Group | Apixaban 2.5mg | Apixaban 5mg | Asprin | Placebo
Started | 165 | 164 | 164 | 164
Completed | 134 | 140 | 143 | 133
Not Completed | 31 | 24 | 21 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban 2.5mg | Apixaban 5mg | Asprin | Placebo | Total
Number analyzed (Participants) | 165 | 164 | 164 | 164 | 657
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 55 [46 to 61] | 52 [47 to 58] | 54 [46 to 59] | 54 [45 to 59] | 52 [46 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 102 | 95 | 96 | 388
  Male | 70 | 62 | 69 | 68 | 269
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 1 | 3
  Asian | 2 | 2 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 0 | 4
  Black or African American | 22 | 20 | 20 | 16 | 78
  White | 124 | 120 | 119 | 131 | 494
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 18 | 22 | 14 | 69
Region of Enrollment [Number; unit: participants]
  United States | 165 | 164 | 164 | 164 | 657

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization for Cardiovascular/Pulmonary Events
Description: The primary outcome will be a composite endpoint of need for hospitalization for cardiovascular/pulmonary events, symptomatic deep venous thrombosis, pulmonary embolism, arterial thromboembolism, myocardial infarction, ischemic stroke, and all-cause mortality for up to 45 days after initiation of assigned treatment.
Time Frame: 45 days
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Apixaban 2.5mg | Apixaban 5mg | Asprin | Placebo
Number analyzed (Participants) | 165 | 164 | 164 | 164
participants | 1 [-2.1 to 4.1] | 1 [-1.5 to 5] | 0 [-0.7 to 10.2] | 0 [-2.7 to 6.8]

ADVERSE EVENTS:
Time Frame: a 45-day treatment period
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Arm/Group | Apixaban 2.5mg | Apixaban 5mg | Asprin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/164 | 0/164 | 0/164
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/164 | 0/164 | 0/164
Other Adverse Events (participants affected / at risk) | 9/165 | 13/164 | 6/164 | 3/164
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 2.5mg (N=165) | Apixaban 5mg (N=164) | Asprin (N=164) | Placebo (N=164)
Non-major Bleeding (Investigations) | 9 | 13 | 6 | 3
Admitted for pneumonia (Reproductive system and breast disorders) | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Early termination leads to a small number of subjects being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT04498273/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT04498273/SAP_002.pdf